CLINICAL TRIAL: NCT01612455
Title: Linking Russian Narcology & HIV Care to Enhance Treatment, Retention, & Outcomes
Brief Title: Linking Infectious and Narcology Care in Russia
Acronym: LINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Samet, Chief, Section of General Internal Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-30414; R01DA032082 (NIH)
Record Dates: First submitted 2012-06-01; First posted 2012-06-05 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: HIV Infection; Drug Use
Keywords: HIV; drug addiction; Russia; case management
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Control participants will receive the narcology hospital's standard of care. With regard to linkage to HIV medical care, patients will be given printed information about where to obtain HIV medical care - the outpatient clinic that is involved in the intervention. Control patients will be referred to outpatient narcology care as part of standard of care. If control participants are newly diagnosed with HIV infection at the addiction hospital, they will receive HIV post test counseling consistent with CDC recommendations (this represents an enhancement of the current standard of care in Russia).
- LINC Case Management (Intervention) (Experimental): LINC Case Management (study Intervention) - see Intervention description
  Interventions: Behavioral: LINC Case Management

INTERVENTIONS:
Behavioral: LINC Case Management — The 1st case management (CM) session will be at the Narcology Hospital and will follow a modified strengths-based case management curriculum. As part of this first session, the CM will show a 10 minute video clip produced by a Russian NGO of HIV-infected patients talking about accessing HIV care. The CM will also tell the patient what his/her CD4 cell count is and discuss what it means with the patient. The case manager will help the client identify the outpatient HIV clinic on a map and will discuss basic drug harm reduction ideas with the client. The remaining 4 CM sessions will happen over the following 6 months. Sessions may happen at the HIV clinic, NGOs, or in the community. The HIV CM helps the client understand the importance of HIV care, identify barriers to care acquisition and recognize one's own strengths, abilities and assets to reduce self-identified barriers to care. The HIV CM's primary aim is to have the client attend an appointment at the HIV outpatient clinic.
  Arms: LINC Case Management (Intervention)

SUMMARY:
The purpose of this study is to implement and assess a behavioral and structural intervention in Russia designed to support and motivate HIV-infected narcology heroin dependent patients (i.e., IDUs) to engage (i.e., initiate and retain) in HIV medical care and ultimately improve their HIV outcomes. The central hypothesis is that an intervention that involves coordination between the narcology and HIV systems via HIV case management delivered by a peer to help motivate and reduce barriers to HIV care will lead to engagement in HIV care.

DETAILED DESCRIPTION:
The objective of this study "Linking Infectious and Narcology Care (LINC)" is to improve upon the treat and retain dimensions of the "seek, test, treat, and retain" paradigm in Eastern Europe. We will implement and assess a behavioral and structural intervention in Russia designed to support and motivate HIV-infected narcology heroin dependent patients (i.e., IDUs) to engage (i.e., initiate and retain) in HIV medical care and ultimately improve their HIV outcomes.

LINC is a clinical model designed to coordinate narcology and HIV systems of care using elements shown to facilitate engagement in medical care: HIV case management and point-of-care CD4 testing. The central hypothesis is that an intervention that involves coordination between the narcology and HIV systems via HIV case management delivered by a peer to help motivate and reduce barriers to HIV care will lead to engagement in HIV care.

Implementation research recognizes that effective interventions may not translate successfully across different contexts and systems. Hence, we will assess the organizational and operational issues that drive engagement in HIV care in Russia.

The project will be undertaken by an international research team experienced in addressing HIV, substance use, and clinical interventions in Russia. This proposal's Specific Aims are to assess the effectiveness of the LINC intervention compared to standard of care on 4 distinct outcomes: 1) initiation of HIV care (> 1 visit to HIV medical care) within 6 months of enrollment; 2) retention in HIV care (> 1 visit to medical care in 2 consecutive 6 month periods) within 12 months; 3) appropriate HIV care (prescribed ART if CD4 cell count is <350 or having a second CD4 count if CD4 ≥350 within 12 months; and 4) improved HIV health outcomes (CD4 cell count at 12 months). The final Specific Aim is to establish the contextual factors that influence adoption and sustainability of the LINC intervention in Russia. If LINC can embed effectively within Eastern European medical systems, then it has the potential to be widely implemented in this region of the world and have a major impact on the HIV epidemic among IDUs.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 70 years
* HIV-infected
* hospitalized at a narcology hospital
* history of injection drug use
* available for CD4 testing
* has 2 contacts to assist with follow-up
* lives within 100 km of St. Petersburg, Russia
* has telephone
* willing to receive care at Botkin Infectious Disease Hospital

Exclusion Criteria:

* currently on ART
* not fluent in Russian
* cognitive impairment precluding informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
1) initiation of HIV care | 6 months
  Greater than or equal to 1 visit to HIV medical care within 6 months of enrollment
2) retention in HIV care | 12 months
  Greater than or equal 1 visit to medical care in 2 consecutive 6 month periods within 12 months
3) appropriate HIV care | 12 months
  prescribed ART if CD4 cell count is less than 350 or having a second CD4 count if CD4 is greater than or equal to 350 within 12 months (Note: As guidelines change over time, this outcome may be updated accordingly.)
4) improved HIV health outcomes | 12 months
  CD4 cell count at 12 months (compared to CD4 cell count at baseline)
5) Establish the contextual factors that influence adoption and sustainability of the LINC intervention in Russia | 4 years
  Qualitative implementation science analysis, including pre-implementation focus groups, interviews, and surveys in Russia; post-implementation qualitative interviews in Russia.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Samet, MD, MA, MPH, Principal Investigator — Boston Medical Center
Locations (3):
- Russia (3):
  - Botkin Infectious Disease Hospital, Saint Petersburg
  - City Addiction Hospital, Saint Petersburg
  - Pavlov State Medical University, Saint Petersburg

REFERENCES:
- [Derived] Gnatienko N, Han SC, Krupitsky E, Blokhina E, Bridden C, Chaisson CE, Cheng DM, Walley AY, Raj A, Samet JH. Linking Infectious and Narcology Care (LINC) in Russia: design, intervention and implementation protocol. Addict Sci Clin Pract. 2016 May 4;11(1):10. doi: 10.1186/s13722-016-0058-5. PMID 27141834